CLINICAL TRIAL: NCT06661304
Title: The Effect of Benson Relaxation Exercise on Anxiety Level and Sleep Quality in Adolescents Receiving Inpatient Treatment in a Psychiatric Clinic: A Randomized Controlled Trial
Brief Title: Effects of Benson Relaxation Exercise on Anxiety Level and Sleep Quality in Adolescents
Acronym: BRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Aydan Akkurt Yalçıntürk, Asst. Prof., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 61351342/020-423
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Relaxation Program; Anxiety; Sleep Quality; Psychiatric Hospitalization
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRE (Experimental)
  Interventions: Other: Benson Relaxation Exercise
- Control (Active Comparator)
  Interventions: Other: Ongoing treatment

INTERVENTIONS:
Other: Benson Relaxation Exercise — Benson relaxation exercise is based on the patient relaxing their body muscles by focusing on deep breathing and a word that means something to them.
  Arms: BRE
Other: Ongoing treatment — In addition to their medical treatment and care in the clinics, patients participate in activities such as group activities, leisure time and walking.
  Arms: Control

SUMMARY:
Purpose: The purpose of this study is to examine the effects of Benson relaxation exercise applied to children and adolescents receiving inpatient treatment in a psychiatric clinic on anxiety levels and sleep quality.

Design: The study is a randomized controlled trial with a pretest-posttest control group.

Method: The study will be conducted in a private psychiatric hospital in Turkey between October 2024 and June 2025. When hospital records were examined, it was determined that 100 patients received inpatient treatment in the last year. Therefore, the universe of the study consisted of 100 patients. The effect of some instructions in the Benson relaxation exercise on delusions and hallucinations is unknown. Therefore, psychosis and schizophrenia patients with delusions and hallucinations will be excluded from the scope of the study. Patients who meet the inclusion criteria will be randomly assigned to the intervention and control groups. The study will be terminated when a total of 60 patients are reached, 30 in the intervention and 30 in the control group. Benson relaxation exercise will be applied to the patients in the intervention group. No application will be made to the patients in the control group. Research data will be collected with the "State-Trait Anxiety Scale" and "Pittsburgh Sleep Quality Index".

Hypotheses:

H1: The anxiety level of patients who applied Benson relaxation exercise is lower than the patients who did not.

H2: The sleep quality of patients who applied Benson relaxation exercise is better than the patients who did not.

ELIGIBILITY:
Inclusion Criteria:

* Being treated in the child and adolescent clinic at the hospital where the study was conducted
* Being between the ages of 14-18
* Not diagnosed with psychotic disorder or schizophrenia
* Scoring between 20 and 59 on the STAI I-II scale
* Scoring 5 and above on the PSQI scale
* Being willing to participate in the study
* Parents giving verbal consent for participation in the study and signing the written voluntary consent form

Exclusion Criteria:

* Not receiving treatment in the child-adolescent clinic at the hospital where the study was conducted
* Not being between the ages of 14-18
* Being diagnosed with psychotic disorder and schizophrenia
* Not receiving a score between 20-59 on the STAI I-II scale
* Receiving a score below 5 on the PSQI scale
* Not being willing to participate in the study
* The parent not giving verbal consent for participation in the study and not signing the written voluntary consent form

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Anxiety Level | Ten days
  State-Trait Anxiety Inventory- STAI I-II. The scale measures anxiety in both healthy and clinical populations. The scale consists of two parts: State Anxiety Inventory (STAI I) and Trait Anxiety Inventory (STAI II). STAI I determines how an individual feels at a certain time and under certain conditions, while STAI II determines how an individual feels regardless of the situation and conditions they are in. Each scale consists of two types of expressions with 20 items. Responses in STAI I and II were assessed on a 4-point scale (not at all, a little, a lot, completely). The total score obtained from both scales ranges from 20 to 80. It has also been shown that people who score higher on STAI scales are more likely to experience anxiety. The Alpha reliability coefficient of the scale was determined to be between 0.94-0.96 for STAI I and 0.83-0.87 for STAI II.
Sleep Quality | Ten days
  Pittsburgh Sleep Quality Index -PSQI: It provides a quantitative measure of sleep quality that is used to define good and bad sleep. PSQI contains a total of 24 questions. 19 of these questions are self-assessment questions. 5 questions are answered by the individual's spouse or a friend. These 5 questions are used only for clinical information and are not included in the evaluation. Self-assessment questions include various factors related to sleep quality. These determine sleep duration, sleep latency (time it takes to fall asleep), and frequency and severity of specific sleep-related problems. The 18 items scored are evaluated with a score between 0 and 3. The sum of the seven component scores gives the total PSQI score. The total score has a value between 0 and 21. A high total scale score indicates poor sleep quality. In the validity and reliability study of the scale, Cronbach's alpha reliability coefficient was found to be 0.80.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar University, Ümraniye, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No